CLINICAL TRIAL: NCT01107171
Title: Multi-center Randomized Controled and Double Blind Trial of Tang-min-ling Pills in the Treatment of Type 2 Diabetes
Brief Title: Trial of Tang-min-ling Pills in the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Tong Xiaolin, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008002P2A02
Record Dates: First submitted 2010-04-15; First posted 2010-04-20 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Tang-min-ling pills;; overweight type 2 diabetes mellitus;; blood glucose; Traditional Chinese Medicine; Clinical Trial; Intervention Studies
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): Tang-min Lin pills analogue
  Interventions: Drug: Placebo
- Tang-min-ling pills high dosage (Experimental): Tang-min-ling pills, high dosage, 12g, tid po
  Interventions: Drug: Tang-min-ling pills high dosage
- Tang-min-ling pills low dosage (Experimental): low dosage group:6g Tang-min-ling pills every time,by 3 times every day for 12 weeks.
  Interventions: Drug: Tang-min-ling pills low dosage

INTERVENTIONS:
Drug: Tang-min-ling pills low dosage — low dosage:6g Tang-min-ling pills every time,by 3 times every day for 12 weeks.
  Other Names: Tang min lin pill
  Arms: Tang-min-ling pills low dosage
Drug: Tang-min-ling pills high dosage — high dosage:12g Tang-min-ling pills every time,by 3 times every day for 12 weeks.
  Other Names: Tang min lin pills
  Arms: Tang-min-ling pills high dosage
Drug: Placebo — Tang-min-Ling pills analogue 6g,tid,po
  Other Names: Tang-min-Ling pills analogue
  Arms: placebo

SUMMARY:
Tang-min-ling pills are made by Chinese herbs extract, and data showed they had antidiabetic effects on the experimental rats and no obvious toxicity was found.This is a randomized, doubled blind, dose-paralleled-control multi-centre clinical trial to evaluate the efficacy and safety of Tang-min-ling pills in the treatment of type 2 diabetic patients and explore the optimal dosage of Tang-min-ling pills.

DETAILED DESCRIPTION:
Two hundred and ten of overweight patients inflicted with primary diabetes mellitus who had stagnated heat of liver and stomach syndrome were recruited, which were randomly divided into 3 groups, and were given high-dosage (12g Tang-min-ling pills every time), low-dosage (6g Tang-min-ling pills every time)、placebo by 3 times every day for 12 weeks respectively. Hemoglobin A1c (HbA1c), Fasting plasma glucose (FPG)、postprandial 2 hours plasma glucose(2hPG)、syndrome、symptoms、body mass index (BMI)、waist circumference (WC) of these groups were measured and analyzed. Some safety indexes such blood and urine and stool routine examination, electrocardiogram (ECG)and liver and kidney function tests were measured and analyzed during the experiment. The treatment period is 12 week.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary type 2 diabetes mellitus
2. BMI ≥ 24 kg•m-2
3. 30-70 years old
4. HbA1c≥7.0%, and FPG>7.0 mmol/L, but <13.9 mmol/L or 2hPG>11.1 mmol/L
5. Informed consent has been signed
6. stagnated heat of liver and stomach syndrome according to TCM syndrome differentiation

Exclusion Criteria:

1. The patients accepted diabetic treatment for more than a month continuously
2. The patients were treated by drugs in 3 week before they were given test drugs
3. Diabetic ketosis, diabetic ketoacidosis or serious inflammation in a month
4. The contractive pressure >160 mmHg or diastolic pressure >100 mmHg
5. Pregnant, preparing for pregnancy or breast-feeding women
6. Mental patients
7. The patients who have serious heart, lung, liver, kidney and brain or other primary complications
8. Allergic persons
9. The patients who are attending other clinical trial
10. The patients who have serious diabetic complications
11. The patients who ever attended this clinical trial
12. Alcohol and / or psychoactive substances, drug abuse and dependency
13. The person maybe loss for some reason such as work or life condition according to the investigator's judgement
14. The lipid-lowering or antihypertensive drug dosage and category which the patients are taking couldn't be kept stable
15. The patients who are eating some drugs or health food which can affect the body weight

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | 12 weeks after treatment
  The HbA1c was measured and analyzed twice, one is before the treatment and the other is 12 weeks aftertreatment to make a self comparison.

SECONDARY OUTCOMES:
Fasting plasma glucose (FPG)、postprandial 2 hours plasma glucose(2hPG)、body mass index (BMI)、waist circumference (WC) | 12 weeks after treatment
symptoms score and Chinese syndrome | 12 weeks after treatment
The rate of adverse events,the blood and urine and stool routine examination, electrocardiogram (ECG)and liver and kidney function tests | 12 weeks after treatment
  The number of participants with adverse events were recorded and compared. The blood and urine and stool routine examination, electrocardiogram (ECG)and liver and kidney function tests were measured and observe the safety.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Tong, Ph.D, Principal Investigator — Guang Anmen Hospital of China Academy of Chinese Medical Sciences
Locations (6):
- China (6):
  - The Affiliated Hospital to Changchun University of Chinese Medicine, Changchun
  - Jilin Hospital of Integrated Traditional and Western Medicine, Changchun
  - Shanghai Shuguang Hospital Affiliated with Shanghai University of Traditional Chinese Medicine, Shanghai
  - The Affiliated Hospital to Liaoning University of Traditional Chinese Medicine, Shenyang
  - The Second Affiliated Hospital to Liaoning University of TCM, Shenyang
  - First Teaching Hospital of Tianjin University of TCM, Tianjin